CLINICAL TRIAL: NCT06840964
Title: Analysis of the Effect of Acidified Omega 3 Esters (DHA+EPA) in Hypertensive Patients With Increased Triglycerides
Brief Title: Effect of Omega 3 in Hypertensive Patients
Acronym: OMECARDIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Maria de la Salud, Argentina (Other)
Collaborators: Gador S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20220325
Record Dates: First submitted 2025-02-11; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; Dyslipidemia
Keywords: hypertension; dyslipidemia; Triglycerides; omega-3 fatty acids
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- O3 Group (Active Comparator): 2 grams/day of omega 3 capsules will be administered orally with food to optimize tolerance. (2 capsules). OMECAP 90 will be used (Registered trademark and approved by ANMAT). The capsules are provided free of charge by the manufacturer. It is recommended not to take on an empty stomach to improve tolerance. It comes in the form of capsules containing 1000 mg of omega 3 ethyl esters at 90%, gelatin 260 mg, glycerin 151 mg and purified water 39 mg.
  Interventions: Dietary Supplement: omega 3 ethyl esters at 90%
- Control Group (Placebo Comparator): Mygliol 812 will be used, a mixture of various medium chain fatty acids (6 to 12 carbon atoms) that are present in various vegetable oils and do not have significant adverse effects. A capsule with the same characteristics as the O3 capsule will be administered and the same administration will be carried out.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: omega 3 ethyl esters at 90% — 2 grams/day of omega 3 capsules will be administered orally, for 12 weeks
  Arms: O3 Group
Dietary Supplement: Placebo — Mygliol 812
  Arms: Control Group

SUMMARY:
This study aims to evaluate the impact of omega-3 (O3) supplementation in participants with high blood pressure and elevated triglycerides, focusing on cardiovascular risk factors. The research is particularly relevant, as O3 has been previously validated for its effects on abnormal lipid levels. The primary and secondary objectives aim to explore the effects of O3, as well as its potential therapeutic benefits in preventing cardiovascular diseases.

The main goal of this research is to investigate how O3 supplementation influences several key cardiovascular risk markers and overall vascular health. Specifically, the study will assess and analyze changes in cholesterol levels, triglycerides, uric acid, and blood glucose levels. Since inflammation plays a major role in heart disease, the study will examine how O3 affects inflammatory markers, including ferritin, high-sensitivity C-reactive protein (hsPCR), and the neutrophil-to-leukocyte ratio. These indicators help determine the level of systemic inflammation in the body. The study also aims to measure whether O3 supplementation improves vascular elasticity.

Apart from the primary cardiovascular effects, the study also aims to determine the tolerance levels of participants receiving O3 supplementation based on their cardiovascular profiles.

The study is based on the hypothesis that taking 2 grams of O3 daily for 12 weeks will lead to a significant reduction in triglyceride levels, lower inflammation markers, improved metabolic risk factors, and enhanced arterial elasticity, which can prevent or slow the progression of cardiovascular diseases. This hypothesis is supported by growing scientific evidence that suggests O3 fatty acids, particularly long-chain polyunsaturated fatty acids (DHA and EPA), have strong cardioprotective properties.

This is a clinical study that is planned in a prospective, interventional, randomized, placebo-controlled, and double-blind format. This means that participants will be randomly assigned to either the treatment group or the placebo group, and neither the participants nor the researchers will know who is receiving the actual treatment until the study ends.

This study is a pilot study, meaning it is a small-scale preliminary study designed to test the hypothesis before conducting a larger trial.

A total of 100 participants will be recruited. Participants will be randomly assigned into two groups: O3 group, receives omega-3 (O3) treatment; and control group, receives a placebo. The assignment will be 1:1 randomization, meaning each participant has an equal (50%) chance of receiving either the treatment or the placebo. The number of participants was chosen based on estimates that a 10% reduction in blood pressure measurements (mean arterial, brachial systolic, brachial diastolic, or central systolic) would be a meaningful outcome.

The duration of omega-3 intervention is based on previous research.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent to participate. Without situations that potentially cause their departure from the country or the possibilities of follow-up during the study.

Diagnosis of hypertriglyceridemia defined as mild 150-199 mg/ moderate 200-499 mg and severe more than 500 mg.

Diagnosis of controlled arterial hypertension (BP ≤140/90 mm Hg) with stable pharmacological treatment (definitions of the Argentine Consensus on HTA, 2018).

Women of childbearing age will be included only if they are under contraceptive treatment, adopted prior to the invitation to participate in the study (hormonal contraceptives (oral, injectable, implantable, etc., intrauterine devices).

Exclusion Criteria:

* Hypersensitivity to the active ingredient, or to soy, or allergy to fish. Liver failure. Pregnancy and breastfeeding. Active anticoagulant treatment. Women of childbearing age who do not use contraceptive methods prior to the invitation to the study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Mean change in office systolic blood pressure from baseline | From enrollment to the end of treatment at 12 weeks
  Mean change in office Systolic blood pressure from baseline in Millimeter Mercury, it measures average changes in office systolic blood pressure.
  Blood pressure is assessed using standardized methods while the participant is seated and resting. The measurement is taken using a validated electronic BP monitor.
Mean change in office diastolic blood pressure from baseline | From enrollment to the end of treatment at 12 weeks
  Mean change in office Diastolic blood pressure from baseline in Millimeter Mercury, it measures average changes in office diastolic blood pressure. Blood pressure is assessed using standardized methods while the participant is seated and resting. The measurement is taken using a validated electronic BP monitor.
Mean change in 24h and Daytime Ambulatory Systolic Arterial Blood Pressure from baseline | From enrollment to the end of treatment at 12 weeks
  Mean change in 24h and Daytime Ambulatory Systolic blood pressure from baseline in Millimeter Mercury, it measures average changes in systolic blood pressure. Blood pressure is assessed using standardized methods for 24 hour ambulatory measurement using a validated BP device monitor.
Mean change in 24h and Daytime Ambulatory Diastolic Arterial Blood Pressure from baseline | From enrollment to the end of treatment at 12 weeks
  Mean change in 24h and Daytime Ambulatory Diastolic blood pressure from baseline in Millimeter Mercury, it measures average changes in diastolic blood pressure. Blood pressure is assessed using standardized methods for 24 hour ambulatory measurement using a validated BP device monitor.
Mean change in resting pulse wave velocity from baseline | From enrollment to the end of treatment at 12 weeks
  Measurement of pulse wave velocity (PWV) in meters per second. The calibrated and validated Mobil-O-Graph® portable monitor (IEM GmbH, Stolberg, Germany) will be used. This module is connected to a computer to record the brachial pulse wave. It performs pulse wave analysis based on the oscillometric method. The arterial pulsation generates pressure oscillations, which are transmitted to the blood pressure cuff and measured by the transducer to be interpreted by a specific software, recording the pulse wave of the brachial artery and deriving a pulse wave from the aortic arch.
  All measurements will be performed on the left arm of the participant, at rest. Subjects will be instructed to be with empty bladder, not to drink coffee 60 minutes before gauging and alcoholic beverage in the last 24 hours.
Mean change in total cholesterol from baseline | From enrollment to the end of treatment at 12 weeks
  Mean change in cholesterol in Milligram/deciliter from baseline, it measures average changes in cholesterol.
Mean change in high density lipoprotein from baseline | From enrollment to the end of treatment at 12 weeks
  Mean change in high density lipoprotein (HDL) in Milligram/deciliter from baseline, it measures average changes in (HDL) cholesterol.
Mean change in triglycerides from baseline | From enrollment to the end of treatment at 12 weeks
  Mean change in triglycerides in Milligram/deciliter from baseline, it measures average changes in plasma triglycerides.
Mean change in fasting blood sugar from baseline | From enrollment to the end of treatment at 12 weeks
  Mean change in fasting blood sugar in Milligram/deciliter from baseline, it measures average changes in fasting blood sugar.
Mean change in high sensitive C reactive protein from baseline | From enrollment to the end of treatment at 12 weeks
  Mean change in high sensitive C reactive protein (Hs-CRP) in Milligram/liter, it measures average changes in high sensitive C reactive protein (Hs-CRP).
Mean change in serum aspartate aminotransferase/serum glutamic-oxaloacetic transaminase from baseline | From enrollment to the end of treatment at 12 weeks
  Serum aspartate aminotransferase/serum glutamic-oxaloacetic transaminase (AST/SGOT) in units per liter (U/L).
Mean change in serum alanine transaminase/Serum Glutamic Pyruvic Transaminase from baseline | From enrollment to the end of treatment at 12 weeks
  Serum alanine transaminase/Serum Glutamic Pyruvic Transaminase (ALT/SGPT) in units per liter (U/L).
Mean change in fasting plasma insulin from baseline | From enrollment to the end of treatment at 12 weeks
  Fasting plasma insulin after fasting for 8-12 hours. Results are reported in micro International Units per milliliter (uIU/mL)
Mean change in serum ferritin from baseline | From enrollment to the end of treatment at 12 weeks
  Serum ferritin is measured in nanograms per milliliter (ng/mL)
Mean change in neutrophil-to-lymphocyte ratio from baseline | From enrollment to the end of treatment at 12 weeks
  The neutrophil-to-lymphocyte ratio (NLR) is a measurement of the number of neutrophils compared to the number of lymphocytes in a blood sample. It's calculated by dividing the absolute neutrophil count by the absolute lymphocyte count. An automated cell counter with mixed technologies performs the calculation.

SECONDARY OUTCOMES:
Tolerability and safety | From enrollment to the end of treatment at 12 weeks
  Presence or not, described by participants, of any of the known side effects , such as belching, indigestion, and diarrhea; or symptoms such as rash, itching, swelling, severe dizziness, or trouble breathing

CONTACTS AND LOCATIONS:
Overall Officials: Virginia C Kotliar, MD, MSc, PhD, Principal Investigator — Santa Maria de la Salud. CONICET
Locations (1):
- Santa Maria de la Salud, San Isidro, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared with the applicant, along with a letter outlining the intended use of the data, which will be submitted to the research board for approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Unending
Access Criteria: A proposal that describes planned analyses must be send by email.